CLINICAL TRIAL: NCT00896922
Title: Assessment of MUM1 Expression, Lymphoma-Associated Macrophages, and Regulatory T-Cells in Follicular Lymphoma: Prognostic Markers in SWOG S8809 and S9800/S9911 Trials Representing Pre-and Post-Monoclonal Antibody Therapy Protocols
Brief Title: S8809-S9800-S9911TM- Biological Markers in Patients With Follicular Lymphoma Treated on Clinical Trial SWOG-8809, SWOG-9800, or SWOG-9911
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000530630; SWOG-S8809/S9800
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Microarray Analysis; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: microarray analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors predict how patients respond to treatment.

PURPOSE: This laboratory study is examining biological markers in patients with follicular lymphoma treated on clinical trial SWOG-8809, SWOG-9800, or SWOG-9911.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the prognostic significance of MUM-1, lymphoma-associated macrophages, and regulatory T cells in patients with follicular lymphoma treated on clinical trials SWOG-8809, SWOG-9800, or SWOG-9911 representing pre- and post-monoclonal antibody therapy protocols.
* Determine whether these factors have similar prognostic significance in patients treated with chemotherapy alone vs chemotherapy and monoclonal antibody therapy on these clinical trials.

OUTLINE: This is a multicenter study.

Previously collected tissue samples from patients are analyzed by immunohistochemistry, gene expression profiling, and quantitative analysis for MUM1 expression, lymphoma-associated macrophages, FOXP3-positive regulatory T cells, CD68, and CD163.

PROJECTED ACCRUAL: A total of 318 samples will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of follicular lymphoma
* Previously treated on any of the following clinical trials:

  * SWOG-8809
  * SWOG-9800
  * SWOG-9911

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled to S8809, S9800 and S9911 consenting to banking
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2007-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Prognostic significance of MUM-1, lymphoma-associated macrophages, and regulatory T cells | Retrospective
Comparison of prognostic significance in patients treated with chemotherapy alone vs chemotherapy and monoclonal antibody therapy | Retrospective

CONTACTS AND LOCATIONS:
Overall Officials: John W. Sweetenham, MD, Study Chair — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: Yes
http://swog.org/Visitors/Download/Policies/Policy43.pdf

REFERENCES:
- [Result] Sweetenham JW, Goldman B, LeBlanc ML, Cook JR, Tubbs RR, Press OW, Maloney DG, Fisher RI, Rimsza LM, Braziel RM, Hsi ED. Prognostic value of regulatory T cells, lymphoma-associated macrophages, and MUM-1 expression in follicular lymphoma treated before and after the introduction of monoclonal antibody therapy: a Southwest Oncology Group Study. Ann Oncol. 2010 Jun;21(6):1196-1202. doi: 10.1093/annonc/mdp460. Epub 2009 Oct 29. PMID 19875761
- [Result] Sweetenham JW, Hsi E, Goldman B, et al.: Numbers of lymphoma associated macrophages (LAMS) and regulatory T-cells (Tregs) in follicular lymphoma (FL) patients (pts) treated with and without monoclonal antibody (MoAb)-containing therapy do not correlate with overall survival (OS): a study from the Southwest Oncology Group (SWOG). [Abstract] Blood 110 (11): A-2602, 2007.